CLINICAL TRIAL: NCT06595888
Title: CT 5400 RT System Application Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300200
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Computed Tomography Workflow Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computed Tomography (Experimental): Human subjects having CT scans
  Interventions: Radiation: Computed Tomography

INTERVENTIONS:
Radiation: Computed Tomography — X-ray by Computed Tomography

SUMMARY:
The purpose of this study is to assess the satisfaction of the common functions, the operation convenience, and the whole system stability, and the safety of CT 5400 RT System.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ Age ≤ 75 years old
* Subjects with Clear consciousness; Subjects can cooperate and act autonomously
* Subjects agree to participate in this clinical study and sign the subject's informed consent
* Women subjects of childbearing age should have a negative pregnancy test and should have no plans to become pregnant in the next 6 months

Exclusion Criteria:

* Subjects who do not have full capacity for civil conduct;
* Women subjects who are pregnant or in lactating phase;
* Subjects who have had a CT scan within one year;
* Subjects with a history of allergies or asthma, severe hepatic and renal insufficiency or hyperthyroidism in which are considered as contraindication for CT contrast-enhanced examination;
* According to the opinion of the investigator: any situation that may affect the evaluation of the results or expose subjects into health risk;
* Subjects with mental disorders who cannot cooperate with the examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
the satisfaction of the common functions | 30 days (anticipated)
  A three-scale assessment will be used for Image exposure level, couch movement, speaker& microphone voice quality, image post processing capability, data storage. A three-scale criteria- Very satisfied, Satisfied, Dissatisfied Assessment criteria: all parameters will be assessed based on the user's feelings. The parameters should all reach "Satisfied", indicating that the general function of the case meet the clinical application requirements.
the operation convenience assessment | 30 days (anticipated)
  A three-scale assessment will be used for laser positioning, panel control, user-friendly interface of post-processing software, operation of post-processing software. A three-scale criteria- Very satisfied, Satisfied, Dissatisfied Assessment criteria: all parameters will be assessed based on the user's feelings. The parameters should all reach "Satisfied", indicating that the general function of the case meet the clinical application requirements.
the system stability assessment | 30 days (anticipated)
  A three-scale assessment will be used for workflow, Image display and transmission, system inactivation, unexpected system shutdown, unexpected termination during scanning, fail to expose during scanning A three-scale criteria- Very satisfied, Satisfied, Dissatisfied Assessment criteria: all parameters will be assessed based on the user's feelings. The parameters should all reach "Satisfied", indicating that the general function of the case meet the clinical application requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China